CLINICAL TRIAL: NCT05195372
Title: The APSANTICO-registry - Evaluation of the Efficacy and Safety of Different Anticoagulants in Patients With Thromboembolic Antiphospholipid Syndrome (APS)
Brief Title: Effectivity and Safety of Different Anticoagulants in Patients With Thromboembolic Antiphospholipid Syndrome
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Other Study IDs: APSANTICO-Registry
Record Dates: First submitted 2021-12-30; First posted 2022-01-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-01

CONDITIONS: Antiphospholipid Syndrome; Venous Thromboembolism; Arterial Thromboembolism; Major Bleed
Keywords: direct oral anticoagulant; vitamin k antagonist; antiphospholipid syndrome; thrombosis; major bleeding
MeSH Terms: conditions — Antiphospholipid Syndrome; Venous Thromboembolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective monocentric registry to evaluate the efficacy and safety of different anticoagulants in patients with thromboembolic antiphospholipid syndrome

DETAILED DESCRIPTION:
Antiphospholipid syndrome is a thrombophilic diathesis characterised by the occurrence of recurrent, unprovoked thromboembolic events (arterial, venous, microvascular) in combination with the presence of specific APS antibodies.

A distinction is made between different subtypes of APS. One is the thrombotic antiphospholipid syndrome (APS), which is the focus of the registry, and the other is obstetric APS, which is characterised by obstetric complications.

The particular challenge in dealing with APS patients is to establish an adequate therapy regime, as some patients suffer from an increased risk of recurrent thrombosis despite anticoagulation and/or aggregation inhibition.

The standard medication for antiphospholipid syndrome is based on the use of vitamin K antagonists (VKA). This regimen is essential to follow, especially in high-risk patients with positive lupus anticoagulants and/or triple positive antiphospholipid antibodies.

In 2019, a 'Red Hand Letter' was issued advising against treating APS patients with direct oral anticoagulants (DOACs) but so far some studies suggest that alternative anticoagulation with DOACs may be beneficial in a selected patient population with a single- or double-positive antiphospholipid antibody profile.

However, the current data on the use of DOAKs in patients with antiphospholipid syndrome is still limited. Therefore, the analysis of the patient data available in the investigator's specialised coagulation centre in the form of the APSantiCO registry should help to select a suitable anticoagulant regimen in everyday clinical practice.

The clinical and laboratory data required for the creation of the register are already available for evaluation in the form of electronic medical records, as the Coagulation Centre of the CCB Bethanien Hospital, which was founded in 2015, has been providing outpatient care to numerous APS patients for years. The data regarding the recording of recurrent thromboses despite anticoagulation and major bleeding under the various anticoagulants are collected with the help of a differentiated study of records. In addition, telephone contact is made with the patients. The telephone contact takes place within the framework of routine quality assurance in order to ensure optimal patient care, since many patients were unable or unwilling to attend their semi-annual or annual routine check-ups in the last two years due to the COVID 19 pandemic situation.

In the course of the telephone call, it should therefore be clarified whether a new appointment is needed, e.g. in case of a new event under the existing medication since the last presentation at the coagulation centre or in case of the occurrence of undesirable side effects and bleeding.

Apart from this telephone call, no patient contact is foreseen.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Confirmed antiphospholipid syndrome with thromboembolic clinical manifestations (VTE, LAE, stroke etc.)
* Patients with APS antibody risk profile (single/double/triple positivity)

Exclusion Criteria:

* APS with isolated pregnancy complications
* No coagulation inhibition
* Inadequately diagnosed APS
* Non-compliance of patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with confirmed thromboembolic antiphospholipid-syndrome who need anticoagulation and/or aggregation inhibition
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Recurrent thromboembolism despite coagulation inhibition | 2015 - 2021
  The main observational variable is the occurrence of recurrent thromboembolic events under DOAC-treatment compared to VKA-treatment and/or other therapeutic regimens (e.g. low molecular weight heparins, aggregation inhibitors) in patients with different APS risk profiles.

SECONDARY OUTCOMES:
major bleeding during coagulation inhibition | 2015 - 2021
  occurrence of major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Principal Investigator — CardioAngiology Center Bethanienhospital (CCB)Frankfurt
Locations (1):
- Edelgard Lindhoff-Last, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No